CLINICAL TRIAL: NCT02345928
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study in Healthy Subjects and Multiple Ascending Dose Study of CNTO 7160 in Subjects With Asthma and Subjects With Atopic Dermatitis
Brief Title: A Single Ascending Dose Study in Healthy Participants and Multiple Ascending Dose Study of CNTO 7160 in Participants With Asthma and Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR105130; CNTO7160ASH1001 (Other: Janssen Research & Development LLC.); 2014-000633-23 (EudraCT Number)
Record Dates: First submitted 2014-08-27; First posted 2015-01-26 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Asthma; Atopic Dermatitis; Healthy
Keywords: Safety; Efficacy; CNTO 7160; Healthy; Asthma; Atopic Dermatitis
MeSH Terms: conditions — Asthma; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (13):
- Part 1: Dose 1 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 1.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 2 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 2.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 3 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 3.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 4 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 4.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 5 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 5.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 6 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 6.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 7 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 7.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 8 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 8.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 1: Dose 9 (Experimental): Drug CNTO7160 or Placebo administered IV infusion Dose 9.
  Interventions: Drug: Part 1: CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 2 (Asthma): Dose 1 (Experimental): Drug CNTO 7160 or Placebo administered IV infusions Dose 1 (3 dose administrations over 4 weeks).
  Interventions: Drug: Part 2 (Asthma): CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 2 (Asthma): Dose 2 (Experimental): Drug CNTO 7160 or Placebo administered IV infusions Dose 2 (3 dose administrations over 4 weeks).
  Interventions: Drug: Part 2 (Asthma): CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 2 (Atopic Dermatitis): Dose 1 (Experimental): Drug CNTO 7160 or Placebo administered IV infusions Dose 1 (3 dose administrations over 4 weeks).
  Interventions: Drug: Part 2 (Atopic Dermatitis): CNTO 7160; Drug: Part 1 and Part 2: Placebo
- Part 2 (Atopic Dermatitis): Dose 2 (Experimental): Drug CNTO 7160 or Placebo administered IV infusions Dose 2 (3 dose administrations over 4 weeks).
  Interventions: Drug: Part 2 (Atopic Dermatitis): CNTO 7160; Drug: Part 1 and Part 2: Placebo

INTERVENTIONS:
Drug: Part 1: CNTO 7160 — Participants will receive Drug CNTO7160 administered IV infusion at escalating doses (with a starting dose of 0.001 mg/kg).
  Arms: Part 1: Dose 1; Part 1: Dose 2; Part 1: Dose 3; Part 1: Dose 4; Part 1: Dose 5; Part 1: Dose 6; Part 1: Dose 7; Part 1: Dose 8; Part 1: Dose 9
Drug: Part 2 (Asthma): CNTO 7160 — Participants will receive Drug CNTO 7160 administered IV infusions (3 dose administrations over 4 weeks).
  Arms: Part 2 (Asthma): Dose 1; Part 2 (Asthma): Dose 2
Drug: Part 2 (Atopic Dermatitis): CNTO 7160 — Participants will receive Drug CNTO 7160 administered IV infusions (3 dose administrations over 4 weeks).
  Arms: Part 2 (Atopic Dermatitis): Dose 1; Part 2 (Atopic Dermatitis): Dose 2
Drug: Part 1 and Part 2: Placebo — Participants will receive single IV infusion of placebo matched to CNTO 7160.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending dose of CNTO 7160 administered intravenously (IV) in healthy participants and multiple dose administered IV in participants with asthma and atopic dermatitis.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, placebo-controlled, multicenter study of CNTO 7160. The study consists of Screening Period, In-patient period (6 days for healthy participants, 11 days for asthmatic participants and atopic dermatitis participants) and outpatient period (105 days for healthy participants, 110 days for asthmatic and atopic dermatitis participants). The total duration of participation for each participant will be approximately 21 weeks for healthy participants, 25 weeks for asthmatic participants, and atopic dermatitis participants. All eligible participants will be randomly assigned to receive active agent or placebo. The study will be conducted in 2 parts. In Part 1, single ascending doses of CNTO 7160 or placebo will be administered to sequential cohorts of healthy participants as an IV infusion. In Part 2, ascending multiple doses of CNTO 7160 or placebo will be administered as IV infusions to sequential cohorts of participants with asthma or atopic dermatitis. Blood samples will be collected for assessment of pharmacokinetic and pharmacodynamics parameters in both part 1 and 2 parameters, along with assessment of safety and clinical effects in part 2. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 (Healthy Participants): Participant must have a body weight in the range of 50 to 100 kilogram (kg) inclusive and have a body mass index (BMI) of 19 to 30 kilogram per meter square (kg/m^2) inclusive
* Part 1 (Healthy Participants): Participant must be healthy on the basis of physical examination, medical history, vital signs and 12-lead ECG performed at screening
* Part 2 (Asthma Participants): Participant must have a body weight in the range of 50 to 125 kg inclusive and have a BMI of 19 to 32 kg/m^2 inclusive
* Part 2 (Asthma Participants): Participant must have a physician documented diagnosis of asthma for at least 12 months before screening
* Part 2 (Atopic Dermatitis Participants): Participant must have a body weight in the range of 50 to 100 kg inclusive and have a BMI of 19 to 30 kg/m^2 inclusive
* Part 2 (Atopic Dermatitis Participants): Participant has physician documented diagnosis of atopic dermatitis for at least 12 months before screening based on UK refinements of the Rajka and Hanifin criteria

Exclusion Criteria:

* Part 1 (Healthy Participants): Participant has any known malignancy or history of malignancy, with the exception of basal cell carcinoma or squamous cell carcinoma in situ of the skin that has been treated with no evidence of recurrence within 6 months prior to the Screening Visit
* Part 1 (Healthy Participants): Participant currently has or has a history of any clinically significant cardiovascular disease, including but not limited to a history of angina or myocardial infarction, congestive heart failure, symptomatic atherosclerotic vascular disease, or arrhythmia.
* Part 2 (Asthma Participants): Participant has any known malignancy or history of malignancy, with the exception of basal cell carcinoma or squamous cell carcinoma in situ of the skin that has been treated with no evidence of recurrence within 6 months prior to the Screening Visit
* Part 2 (Asthma Participants): Participant has or have had a serious infection (eg, sepsis, pneumonia or pyelonephritis), or have been hospitalized or received IV antibiotics for a serious infection during the 4 months prior to the Screening Visit
* Part 2 (Atopic Dermatitis Participants): Participant has any known malignancy or history of malignancy, with the exception of basal cell carcinoma or squamous cell carcinoma in situ of the skin that has been treated with no evidence of recurrence within 6 months prior to the Screening Visit.
* Part 2 (Atopic Dermatitis Participants): Participant has or have had a serious infection (eg, sepsis, pneumonia or pyelonephritis), or have been hospitalized or received IV antibiotics for a serious infection during the 4 months prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability of CNTO 7160 (Part 1) | Through Week 17
  The incidence of TEAEs from treatment until the last scheduled follow-up visit will be summarized by treatment group.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability of CNTO 7160 (Part 2) | Through Week 21
  The incidence of TEAEs from treatment until the last scheduled follow-up visit will be summarized by treatment group.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) (Part 1) | Up to Week 17 after dose
  Cmax (microgram per millileter [mcg/mL]) will be summarized by treatment group.
Maximum Observed Serum Concentration (Cmax) (Part 2) | Up to Week 21 after dose
  Cmax (mcg/mL) after the first and last dose will be summarized by treatment group.
Area Under the Serum Time Curve [AUC(0-t) and AUC(0-infinity)] (Part 1) | Up to Week 17 after dose
  AUC (mcg*day/mL) will be summarized by treatment group.
Area Under the Serum Concentration Versus Time Curve [AUC(t1-t2)] (Part 2) | Up to Week 21 after dose
  AUC (mcg*day/mL) will be summarized by treatment group.
Number of Participants With Antibodies to CNTO 7160 (Part 1) | Up to Week 17
  The incidence of participants with anti-CNTO 7160 antibodies will be summarized by treatment group.
Number of Participants with Antibodies to CNTO 7160 (Part 2) | Up to Week 21
  The incidence of participants with anti-CNTO 7160 antibodies will be summarized by treatment group.
Change From Baseline in Immunoglobulin E (IgE) (Part 2) | Baseline, Week 21
  Change from Baseline in immunoglobulin E (IgE) Concentration (international unit per millileter [IU/mL]) through Week 21 will be summarized by treatment group.
Change from Baseline in Chemokine (C-C motif) Ligand 17 (CCL17) (Part 2) | Baseline, Week 21
  Change from Baseline in Chemokine (C-C motif) Ligand 17 (CCL17) concentration (picogram per millileter [pg/mL]) through Week 21 will be summarized by treatment group.
Change From Baseline in Forced Expiratory Volume in 1 second (FEV1) in Participants With Asthma | Baseline Up to week 21
  Changes in FEV1 (liter [L]) from baseline through end of follow up will be summarized by treatment group.
Change From Baseline in Eczema Area Severity Index (EASI) in Participants With Atopic Dermatitis | Baseline up to week 21
  Changes in EASI score from baseline through the end of follow up will be summarized by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- Belgium (2):
  - Antwerp
  - Merksem
- Germany (5):
  - Berlin
  - Hamburg
  - Hanover
  - Kiel
  - Mönchengladbach

REFERENCES:
- [Result] Nnane I, Frederick B, Yao Z, Raible D, Shu C, Badorrek P, van den Boer M, Branigan P, Duffy K, Baribaud F, Fink D, Yang TY, Xu Z. The first-in-human study of CNTO 7160, an anti-interleukin-33 receptor monoclonal antibody, in healthy subjects and patients with asthma or atopic dermatitis. Br J Clin Pharmacol. 2020 Dec;86(12):2507-2518. doi: 10.1111/bcp.14361. Epub 2020 Jun 14. PMID 32415720